CLINICAL TRIAL: NCT03499366
Title: A Clinical Observational Follow-up Study of European Pediatric Cases of Acute Flaccid Myelitis Associated With EV-D68 Infection.
Brief Title: European Paediatric AFM Associated With EV-D68 Follow-up Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University Medical Center Groningen (Other); National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Helle Cecilie Viekilde Pfeiffer, Researcher, Pricipal investigator, PhD, Department of Child Neurology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/2123
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Flaccid Hemiplegia; Flaccid Paraplegia; Flaccid Tetraplegia, Unspecified; Enterovirus D68; Myelitis, Infectious
Keywords: enterovirus D68; AFP; AFM; EV-D68; acute flaccid myelitis; acute flaccid paresis
MeSH Terms: conditions — Hemiplegia; Paraplegia; Quadriplegia; Myelitis; acute flaccid myelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HFMS, MRC, ACTIVLIM, PedsQl-4.0 — Clinical performance tests, quality of life, activity of daily life form.

SUMMARY:
The study is a follow-up study on children with acute flaccid paresis associated with enterovirus D68 infection. Only children living in Europe are eligible. The study aim is to clarify the outcome of the disease and investigate possible clinical correlation with outcome, including initial severity, demographic characteristics, treatment and MRI findings.

DETAILED DESCRIPTION:
Title: Clinical observational follow-up study of children with Acute Flaccid Myelitis associated with EV-D68 infection- a cross European collaboration.

Study objectives: To study the clinical outcome and function of patients with Acute Flaccid Myelitis associated with enterovirus (EV)-D68 infection after 1 to 3 years, in order to assist clinicians in providing prognoses for patients and to guide further investigation.

Primary objective will be:

• Functional assessment using the Hammersmith Functional Motor Scale (HFMS) -score at follow up; 1, 2 and three years depending on time of debut

Secondary objectives are to describe these secondary outcomes and their changes over time, from onset to 1, 2 and 3 years, depending on time of debut:

* Medical Research Council (MRC) sum score at acute illness and at 1, 2 and 3 years follow up depending on time of debut as well as possible improvements over time
* MRC score in the most affected joint at acute illness and at 1, 2 and 3 years follow up depending on time of debut, as well as possible improvements over time ACTIVLIM functional score at 1, 2 and 3 years follow up depending on time of debut
* Quality of life at 1, 2 and 3 years follow up depending on time of onset measured using the Paediatric Quality of Life Inventory (PedsQL) 4.0.
* Number of days needing intensive care (range and mean)
* Number of days needing mechanical ventilation (range and mean)
* Number of deaths will be reported
* Number of complete recoveries will be reported

Explorative objectives:

* Exploring demographic parameters and how it relates to outcome (HFMS/ MRC-score/ ACTIVLIM/ PedsQL 4.0)
* Exploring different treatments and how it relates to outcome (HFMS/ MRC-score/ ACTIVLIM/ PedsQL 4.0)
* Exploring different clinical parameters and how it relates to outcome (HFMS/ MRC-score/ ACTIVLIM/ PedsQL 4.0)
* Exploring time aspects of the recovery process (individual MRC-score and MRC sum score changes).
* Characteristics on MRI will be explored with regards to outcome measures (HFMS/ MRC-score/ ACTIVLIM/ PedsQL 4.0)
* In cases with repeated MRI scans, changes will be described
* In cases with repeated neurophysiological examinations, changes will be described.

Clinical study/intervention design: This is a clinical observational study aiming at including all registered European AFM-EVD68 patients less than 18 years of age.

Safety endpoints: There is no treatment given in this study. If we become aware of important safety issues concerning included patient's treatment regimens or supportive treatment the responsible treating physician well be informed promptly via e-mail.

Duration of study: The study is intended to produce follow up data every year for two years. Inclusion will begin in March 2018 and the study terminates in March 2020. Analysis of data might hereafter continue for one year.

Follow-up: The study is a follow up study itself. Follow up will be done as close to 1 year after onset as possible and hereafter every year for minimal 2 years.

The study is intended as a clinical follow-up study exploring the outcome of patients with acute flaccid paresis associated with enterovirus D68. The patients will undergo a standard neurologic examination and assessment using Hammersmith functional motor scale expanded. The parents/ child will be asked to fill out a form concerning quality of life and activity of daily living. There will be no painful or invasive procedures and the duration of each visit can be expected to be approx. 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Acute flaccid paresis (AFP) at onset, and
* Enterovirus D-68 polymerase chain reaction (PCR) positive in any specimen in a timely sample (+/- 3 weeks from onset of paresis), and
* Age <18 years at onset, and
* Magnetic resonance imaging (MRI) of spine and brain at onset with signs of myelitis.

Exclusion Criteria:

* Major trauma
* central nervous system (CNS) malignancy
* Bleeding or infarctions in CNS
* Previous demyelinating disease
* Other infections cause of myelitis is more likely
* Patient and/or legal guardian is not able/willing to sign the consent form

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-04-09 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Total Hammersmith Functional Motor scale- score at follow-up | 1 year
  O'Hagen, J. M., et al. (2007). "An expanded version of the Hammersmith Functional Motor Scale for SMA II and III patients." Neuromuscul Disord 17(9-10): 693-697.Neurol. 2003;7(4):155-9.
  The scale is a 33 items evaluation (0, 1 or 2 points in each item) and results in an overall functional score. Range: 0-66, with a higher score reflecting better performance. No sub-scores will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Anette ramm-Pettersen, MD, PhD, Study Chair — Head of department
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided